CLINICAL TRIAL: NCT06756711
Title: Combination of Supplements for Treating Autistic Spectrum Disorder
Acronym: APITSA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundatia Bio-Forum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BF-045
Record Dates: First submitted 2024-12-23; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder (ASD
Keywords: Autistic Spectrum Disorder; apitherapy; brain aromatase
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Plant Extracts

STUDY DESIGN:
Intervention Model Description: prospective, double-blind, placebo-controlled, crossover, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active combination (Active Comparator): A combination of 3 supplements with royal jelly and various plant extracts
  Interventions: Dietary Supplement: A combination of apitherapy and plant extracts
- Placebo combination (Placebo Comparator): A combination of 3 products with identical look and colour
  Interventions: Combination Product: Placebo Combination

INTERVENTIONS:
Dietary Supplement: A combination of apitherapy and plant extracts — This combination contains the active comparator
  Arms: Active combination
Combination Product: Placebo Combination — A combination containing inert substances - placebo
  Arms: Placebo combination

SUMMARY:
A pilot study to compare the efficacy of a combination of apitherapy supplements versus placebo in children with autistic spectrum disorder.

DETAILED DESCRIPTION:
A prospective, double-blind, placebo-controlled, crossover, multicentre clinical study which will enrol up to 45 children diagnosed with ASD (enrolment will stop when 40 children have completed the study). Children ages 3-14 will be tested before and after administering the combination of active substances (3 months) and placebo (3 months). The duration of participation in the study for each child will be 6 months. The supplements tested consist of three products - a combination of apitherapy and plant extracts - which have been approved for sale as individual supplements for more than 5 years in Romania - Apicol 12 gamma, Laptisor de matca activat (Royal Jelly) and Telom R Cerebral. Participation in the study is free and all children will be comparatively evaluated with the ATEC and ASRS scales and three sets of blood tests.

ELIGIBILITY:
Inclusion Criteria:

* age 3-14 years
* diagnosed with typical or atypical autism spectrum disorder (F84.0 or F84.1) and received at least one therapeutic intervention before enrolling
* the ability to follow an oral treatment, with TID/BID/QD administration
* the availability to perform 3 sets of blood tests at a clinical laboratory within 6 months (initial, at 3- and 6-months)
* the availability to perform 3 visits to the Investigator and 3 psychometric evaluations within 6 months

Exclusion Criteria:

* patients enrolled in another interventional clinical trial currently or which ended less than 1 month prior to enrolling in this study
* known allergy to hive products or one of the substances studied
* inability to perform the study requirements (3 visits to the Investigator, 3 psychometric assessments, 3 sets of blood tests)
* diagnosis of diabetes
* history of seizures/epilepsy
* administration of anticoagulants, antiplatelets, thrombolytic agents, low molecular weight heparins, anticonvulsants, insulin, monoamine oxidase inhibitors, non-steroidal anti-inflammatory drugs or thiazide diuretics
* allergy to celery and other plants of the Fam. Apiaceaea (Umbelliferae)
* abnormally elevated baseline (at V1) values of ferritin, homocysteine, HgbA1c, ESR

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Modification on ATEC score | 3 months each of administration of active treatment and respectively placebo
  Total ATEC (Autism Treatment Evaluation Checklist) scores before and after each intervention, as well subscale scores; higher scores indicate worse status, score range between 0 (minimal, absence of pathology), to 180 - maximal intensity of symptoms
Modification of ASRS scores | 3 months each of administration of active treatment and respectively placebo
  Scores on Autism Spectrum Rating Scales (ASRS) tests, total and 8 subscales will be compared before and after each intervention; total scores vary between 50-255, with higher score indicating more severe symptoms

SECONDARY OUTCOMES:
NSE level modifications | 3 months each of administration of active treatment and respectively placebo
  Changes in the levels of serum Neuron-specific enolase (NSE) will be compared between the two arms, higher levels indicate higher neuronal destruction

OTHER OUTCOMES:
Adverse effects | 3 months each of administration of active treatment and respectively placebo
  Adverse effects will be noted and compared for the two study arms

CONTACTS AND LOCATIONS:
Overall Officials: Felician Stancioiu, M.D., Principal Investigator — Fundatia Bio-Forum
Locations (2):
- Romania (2):
  - Clinica Aide Sante, Bucharest
  - Medical Link SRL, Constanța

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stancioiu F, Bogdan R, Dumitrescu R. Neuron-Specific Enolase (NSE) as a Biomarker for Autistic Spectrum Disease (ASD). Life (Basel). 2023 Aug 13;13(8):1736. doi: 10.3390/life13081736. PMID 37629593

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT06756711/Prot_SAP_ICF_000.pdf